CLINICAL TRIAL: NCT06496347
Title: CBB Satisfaction Survey
Status: Completed | Type: Observational
Sponsor: Cheng Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Cheng Sheng Chen, Director, Department of Psychiatry, Kaohsiung Medical University
Organization: Kaohsiung Medical University (Other)
Other Study IDs: CBB-TWSS-21
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy control (HC) group,: no intervention(s)
- MCI/dementia group: no intervention(s)

SUMMARY:
The Cogstate Brief Battery (CBB) is a computerized measure for cognitive screening that consists of four cognitive tasks to assess psychomotor function, attention, learning, and working memory, and provides an easy-to-interpret report without the need for manual scoring. Clinical trials and research studies have proven the validity of CBB for cognitive assessment and distinguish MCI or dementia from normal aging.

Participants express a growing acceptance of the use of computerized tests for detecting cognitive impairment, viewing it as a potential tool to improve quality of patient care and the patient-clinician relationship when used in conjunction with the "human touch." The CBB utilizes non-verbal playing-card stimuli in order to minimize language, educational and cultural biases affecting performance. It has the advantages of being portable (adaptable to notebooks, tablets, and even smart phones), short (20-30 min), game-like in presentation and thus motivating, and cross-culturally adaptable. The CBB is well liked in waiting rooms of primary care settings. It is assumed that the CBB will also be highly accepted by Taiwanese.

ELIGIBILITY:
For MCI/dementia groups:

Inclusion criteria:

1. Patient diagnosed with MCI, AD dementia, VaD or DLB
2. Participant who is 50-85 years of age
3. Taiwanese who had finished primary education
4. Participant (or legally acceptable representative) who signed the written ICF

Exclusion criteria:

1. Participant with GDS score ≥ 10
2. Participant with CDR score > 1 (Assessment result within 6 months can be used conditionally.)
3. Participant with MMSE score ≤ 17 (MMSE score will be converted from CASI score. Assessment result within 6 months can be used conditionally.)
4. Participant diagnosed with Schizophrenia
5. Participant diagnosed with Parkinson's disease
6. Participant diagnosed with cancer (except basal cell skin carcinoma) in the past two years
7. Participant diagnosed with uncontrolled diabetes
8. Participant with regular alcohol use exceeding two standard drinks per day for women or four per day for men (one standard drink corresponds to 350 cc of beer)
9. Participant unable to take CBB test according to the investigator's discretion, such as blindness
10. Participant who, in the opinion of the investigator or medical monitor, should not participate in the study

For HC group:

Inclusion criteria:

1. Healthy volunteers without objective cognitive impairment
2. Participant who is 50-85 years of age
3. Taiwanese who had finished primary education
4. Participant who signed the written ICF

Exclusion criteria:

1. Participant with GDS score ≥ 10
2. Participant diagnosed with Schizophrenia
3. Participant diagnosed with Parkinson's disease
4. Participant diagnosed with cancer (except basal cell skin carcinoma) in the past two years
5. Participant diagnosed with uncontrolled diabetes
6. Participant with regular alcohol use exceeding two standard drinks per day for women or four per day for men (one standard drink corresponds to 350 cc of beer)
7. Participant unable to take CBB test according to the investigator's discretion, such as blindness
8. Participant who, in the opinion of the investigator or medical monitor, should not participate in the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two hundred seventy-one participants are planned to be recruited and it is expected to have 180 eligible participants for data analysis with 33% dropout rates estimated. The distribution of the number of participants is as follows:
  Participant group estimate enrolled participant no. eligible participant no. HC (healthy control) 60 40 MCI 60 40 AD 75 50 VaD 38 25 DLB 38 25
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
CBB Testing Score and Brain Age Score | Data analysis and study report: 3 months
  Participant satisfaction with using CBB will be measured by the paper-and-pencil satisfaction survey including 15 questions. See Appendix 1: Satisfaction Survey for Participant. Score of Question 2 will be ranged from "Strongly agree" (1) to "Strongly disagree" (5). Scores of Question 3~13 will be ranged from "Strongly disagree" (1) to "Strongly agree" (5).
  The participant satisfaction rates will be estimated from Question 2, 3, 5, 6, 8, 9, 11, 12 and 13, and calculated in accordance with the following formula:
  Satisfaction rate = (number of score 5 and 4 / number of answers) x 100% The satisfaction rate of each question mentioned above and the frequency of each score of each question will be evaluated and presented by groups of HC and MCI.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes